CLINICAL TRIAL: NCT01184352
Title: Registry for PCI With the TriReme Medical, Inc. Glider(TM) PTCA Balloon Catheter
Brief Title: Glider PTCA Balloon Catheter Registry
Status: Completed | Type: Observational
Sponsor: TriReme Medical, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CLR734
Record Dates: First submitted 2010-08-16; First posted 2010-08-18 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PCI patients treated with Glider Device
  Interventions: Device: TriReme Medical, Inc. Glider(TM) PTCA Balloon Catheter

INTERVENTIONS:
Device: TriReme Medical, Inc. Glider(TM) PTCA Balloon Catheter — Percutaneous Coronary Interventions performed with the Glider PTCA Balloon Catheter

SUMMARY:
The objective of this Registry is to demonstrate the utility of the Glider PTCA Balloon Catheter for crossing during the treatment of coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing PCI who are at least 18 years old
* PCI procedure included the use of at least one Glider PTCA Balloon Catheter
* Patient has been informed, in accordance with local requirements, that their data will be used in the Glider Registry

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated by Physicians using the Glider PTCA Balloon Catheter who are willing to participate in the Glider Registry.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2010-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Technical Success | average of 1 hour
  Percentage of lesions successfully crossed among those attempted with the Glider PTCA Balloon Catheter as assesed during procedure.

SECONDARY OUTCOMES:
Procedure Success | average of 2 days
  Percentage of patients treated with at least one Glider PTCA Balloon Catheter having <50% residual diameter stenosis, or TIMI 3 flow if at a bifurcation side branch, without the development of in-hospital MACE (Major Adverse Cardiac Event).

CONTACTS AND LOCATIONS:
Overall Officials: Carlo DiMario, MD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (6):
- Germany (5):
  - Vivantes Klinikum Zum Friedrichshain, Berlin
  - Klinikum Coburg Herzkatheterlabor, Coburg
  - Alfried Krupp Khs, Essen
  - Elisabeth-Krankenhaus Essen Kardiologie, Essen
  - University Klinikum Muenster, Münster
- Royal Brompton Hospital, London, United Kingdom